CLINICAL TRIAL: NCT03873831
Title: Clinical Trial of the Effects of Therapy Dogs on Social Behavior in Group Social Skills Instruction With Children With Autism
Brief Title: Effects of Therapy Dogs on Social Behavior in Group Social Skills Instruction With Children With Autism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Texas Tech University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, CassiDe Street, Director, HRPP, Texas Tech University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: Therapy Dogs Group Autism; R21HD095206 (NIH)
Record Dates: First submitted 2019-03-06; First posted 2019-03-14 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Autism Spectrum Disorder; Social Skills
Keywords: Therapy dog; Autism Spectrum Disorder; Social skills; Group therapy
MeSH Terms: conditions — Autism Spectrum Disorder; Social Skills

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Social Skills Control (A-A) (Active Comparator): The children in the "A-A" condition, a true control, will remain without a dog for the full 10 weeks.
  Interventions: Behavioral: Social skills group
- Social Skills Dog (A-B) (Experimental): The "A-B" condition will involve standard instruction for 5 weeks ("A"), followed by 5 weeks of group instruction while a therapy dog is present in the room ("B").
  Interventions: Behavioral: Animal-assisted intervention; Behavioral: Social skills group
- Social Skills Dog (B-A) (Experimental): The "B-A" condition will be identical, except the first 5 weeks of instruction will include the dog, followed by 5 weeks of standard instruction with no dog.
  Interventions: Behavioral: Animal-assisted intervention; Behavioral: Social skills group

INTERVENTIONS:
Behavioral: Animal-assisted intervention — The therapy dog is present during the session.
  Other Names: Therapy dog
  Arms: Social Skills Dog (A-B); Social Skills Dog (B-A)
Behavioral: Social skills group — The group program is 10 weeks in duration, with 1-hour long sessions once per week. Children will be taught new social skills each week using an established teaching interaction procedure, in which the therapist first describes the target skill, provides a rational and context for the behavior, divides the skill into smaller steps, demonstrates the behavior, and has each learner role-play the skill while providing feedback in the form of praise and tokens and corrective instruction. The last week involves a probe "free-play" session, in which children are assessed in a more naturalistic environment without any corrective feedback from therapists.

SUMMARY:
Animal-Assisted Interventions (AAI) can increase social behavior in children with autism spectrum disorder (ASD), although the mechanism by which this occurs remains elusive. The central goal of this project is to identify the mechanisms involved in the social-enhancing effect of dogs on children with ASD. The investigators will incorporate therapy dogs into an established evidence-based, group social skills instruction program for children with ASD, using a controlled experimental design with between- and within- subject comparisons and physiological and behavioral outcome measures. The investigators predict therapy dogs to have a specific and measurable effect on children's social behavior and that this effect is gained through identifiable mechanisms. Specifically, the investigators hypothesize that (1) an integration of therapy dogs into group social skills instruction will result in reduced stress and improved social behavior compare to traditional group instruction; (2) repeated exposure to the therapy dog across sessions will increase a child's preference for spending time with the dog and will increase the social-enhancing effects of the dog; and (3) that the therapists will experience less stress, engage in more social and affiliative behavior towards the children, and deliver higher quality instruction during sessions that include dogs. The investigators will enroll 72 children with ASD into group social skills instruction classes taught by 6 therapists. Each child will experience a 10-week, 8-student class in which either (a) the first 5 weeks will involve a therapy dog, (b) the last 5 weeks will involve the therapy dog, or (c) the class will not involve a therapy dog. The therapists will teach the courses repeatedly across the three cycles of the program with different children, rotating through each condition. Social behavior, stress behavior, heart rate, electrodermal activity, and salivary cortisol concentrations of children and therapists will be assessed and compared across conditions. The direction of the children's social behavior towards the dog and peers and the changes in quality of instruction of therapists during dog sessions compared to no-dog sessions will also be assessed. The outcomes of this research will lead to significant enhancements in current interventions for individuals with ASD.

DETAILED DESCRIPTION:
Approximately 1 in 68 children are diagnosed with autism spectrum disorder (ASD). The most detrimental hallmarks of autism are significant deficits in social and conversational skills, resulting in difficulties forming and maintaining social relationships. Children who have few friends are at a high risk for having depression, doing poorly in school, and not being employed as adults. Animal-Assisted Interventions (AAI) have been shown to increase social behavior in both children with ASD as well as in various human populations. Children with ASD display more social behavior in a classroom setting when a therapy dog is present, but while the effect dogs have on increasing social behavior has been well-established, the mechanism by which this increase occurs remains elusive.

Our long-term goal is to identify causal mechanisms that may ameliorate the social behavior deficit in autism. The specific goal of this research is to identify the mechanisms involved in the social-enhancing effect of dogs on children with ASD. Our central hypothesis is that therapy dogs have a specific and measurable effect on children's social behaviors. Furthermore, by directly testing a number of significant confounds frequently found in AAI research (novelty effects and the effects of the dog on the therapist), the investigators will rule out alternative hypotheses. It has been suggested that the effects of AAI are partly caused by the novelty of having an animal in a location where animals are not typically seen (such as a classroom) rather than caused by an underlying feature specific to the animal. Additionally, the therapist's potentially altered quality of instruction in response to the presence of a dog in the room has not been previously explored.

The investigators will attain our goal by incorporating therapy dogs into an established group social skills instruction program for children with ASD, using a quasi-experimental, repeated-measures counter-balanced mixed design with physiological and behavioral outcome measures. Furthermore, using a rigorous experimental single-subject design, the investigators will assess the effect of the dogs on therapists. Group social skills instruction interventions based on the principles of applied behavior analysis (ABA) and that target conversational and communication skills have been shown as particularly successful at improving social behavior in individuals with ASD. Despite the beneficial outcomes, any educational interventions, especially those that require social interaction, can be a source of stress for children with ASD, and stress can impact learning and memory. Creating an educational setting that balances the levels of stress is beneficial. Dogs may have a stress-ameliorating effect on the child, thereby allowing social behavior to emerge during the instructional period and enhance the child's ability to learn social skills. Another barrier to effective instruction may be that peer-to-peer contact is perceived as highly aversive to children with ASD. Thus, by providing a non-judgmental therapy dog learning partner, the children may first practice social skills in a safer environment, free from negative feedback.

Aim 1: Identify the mechanism by which dogs increase group social behavior in children with ASD.

The investigators will directly test two complementary hypotheses: (1) stress-ameliorating effect of the dog on the child, and (2) the dog as a non-judgmental learning partner. The investigators predict that the presence of the dog in group social skills instruction program (n = 72 children, with 8 children per group) will not only improve the quantity and quality of social behavior, but also reduce physiological (salivary cortisol, heart rate, and electrodermal activity) and behavioral signs of stress compared to the absence of the dog. The investigators further predict that during therapy sessions with dogs, most of the children's social behavior will be directed towards the dog rather than peers.

Aim 2: Identify if and how repeated exposure to the dog influences social behavior of children with ASD.

The investigators hypothesize that repeated exposure to the therapy dog across sessions will alter 1) the preference to spend time with the dog, as measured by changes in time spent in proximity, and 2) the social-enhancing effects of the dog.

Aim 3: Identify the effects of the dog on the therapist. The investigators hypothesize that during repeated sessions with the dog, therapists (n = 6) will experience less stress (as measured by salivary cortisol, heart rate, and electrodermal activity), engage in more social and affiliative behavior towards the children, and deliver higher quality instruction.

The outcomes of this research will lead to significant enhancements in the current understanding of the mechanism by which dogs increase social behavior in children with ASD.

The innovative combination of methodologies from animal science and ABA therapy is uniquely suited for the determination of the mechanism of the social-enhancement effect of dogs. By measuring both behavioral responses and physiological biomarkers of stress during the intervention, the investigators will determine the mechanism through a rigorous and all-inclusive approach. Furthermore, by directly assessing two key confounding variables, the novelty effect and the effect of the dog on the therapist, the investigators will pave the way for more rigorous research into AAI. Completion of this research will expand our knowledge about the mechanism by which dogs may benefit children with ASD, introduce new intervention methods to provide longer-term benefits for children, and provide a starting point for research into new interdisciplinary technology using animals in ABA-based therapy.

ELIGIBILITY:
Inclusion Criteria:

* Children 11-17 years of age
* Children with a diagnosis of autism spectrum disorder (ASD)
* Children with receptive and expressive language skills

Exclusion Criteria:

* Foster children
* Children with a phobia of dogs as reported by a parent or any behavioral signs during the study (crying, withdrawing from dog, body shaking, verbal report, etc.)
* Children with a history of animal mistreatment, abuse, or aggressive behavior toward animals as reported verbally by parents and/or through the screening questionnaire (Children's Attitude and Behaviors towards Animals, CABTA), or any behavioral signs (attempts to swat, hit, pinch, kick or pull the dog's hair) during the study
* Children who have a service animal as reported by the parent

Ages: 11 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 72 (Actual)
Dates: Start 2019-05-15 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-04-26 (Actual)

PRIMARY OUTCOMES:
Verbal utterances | Sessions 1 through 10 (duration of 10 weeks)
  The investigators will record total frequency and rate of verbal utterances during each session.
Direction of utterances | Sessions 1 through 10 (duration of 10 weeks)
  The investigators will record the direction of the utterance: towards peers, the therapist, or the therapy dog.
Quality of utterance | Sessions 1 through 10 (duration of 10 weeks)
  The investigators will record the quality of the utterances (e.g., rude and friendly words, greetings, etc.).
Unwanted behavior | Sessions 1 through 10 (duration of 10 weeks)
  Data on the presence of anxious or problem behavior (e.g., tantrum, non-compliance, crying, stereotypy) will be collected using a partial-interval coding with 5-s time bins method.
Social behavior | Sessions 1 through 10 (duration of 10 weeks)
  Data on the presence of social behavior (e.g., smiling, proximity to others, speaking) will be collected using a partial-interval coding with 5-s time bins method.
Heart Rate | Sessions 1 through 10 (duration of 10 weeks)
  To obtain a continuous measure heart rate, the investigators will use a NeuroLynQ Galvanic Skin Response (GSR) unit (Shimmer, Boston, MA), which uses phasic conductance and an optical pulse sensing probe. The small portable wristband device attaches to three sensors that are placed on the fingers of the non-dominant hand using Velcro straps. The device is lightweight and comfortable. These devices will be placed on each student and therapist at the beginning of each session and removed at the end of each session. The data from the devices will be collected at the end of each session.
Electrodermal activity | Sessions 1 through 10 (duration of 10 weeks)
  To obtain a continuous measure of electrodermal activity, the investigators will use a NeuroLynQ Galvanic Skin Response (GSR) unit (Shimmer, Boston, MA), which uses phasic conductance and an optical pulse sensing probe. The small portable wristband device attaches to three sensors that are placed on the fingers of the non-dominant hand using Velcro straps. The device is lightweight and comfortable. These devices will be placed on each student and therapist at the beginning of each session and removed at the end of each session. The data from the devices will be collected at the end of each session.
Salivary cortisol | Sessions 1 through 10 (duration of 10 weeks)
  At the beginning and/or the end of the session, each child and therapist will be asked to provide a saliva sample. The saliva collection procedures are based on established practices with children and will involve placing a cotton swab Salimetrics Child Swab) into the child's mouth for 1 min.

SECONDARY OUTCOMES:
Quality of instruction: correct and timely feedback | Maximum of 50 weeks
  The quality of instruction will be measured by trained observers through the proportion of correct and timely feedback given to the children.
Quality of instruction: adherence to the program script | Maximum of 50 weeks
  The quality of instruction will be measured by trained observers by marking the level of adherence to the program script.
Quality of instruction: attention to children | Maximum of 50 weeks
  The quality of instruction will be measured by trained observers by recording the level of attention provided for each child.

CONTACTS AND LOCATIONS:
Overall Officials: Wesley H Dotson, PhD, BCBA-D, Principal Investigator — Texas Tech University
Locations (1):
- Texas Tech University, Lubbock, Texas, United States

IPD SHARING:
Plan to Share IPD: No
The researchers are committed to sharing research data according to the most recent NIH guidelines (https://grants.nih.gov/grants/policy/data_sharing/), while also understanding our duty to protect the privacy of our research participants. De-identified data will be shared among PIs through OneDrive, a secure university web-based application.